CLINICAL TRIAL: NCT03343236
Title: Inflammation and Metabolism After Radiotherapy- Predictors of Survival in Patients with Head and Neck Cancer
Brief Title: Nutrition and Inflammation in Patients with Head and Neck Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Swedish Cancer Society (Other); The Kamprad Family Foundation for Entrepreneurship, Research & Charity (Other); AFA Insurance (Industry)
Responsible Party: Sponsor
Other Study IDs: 160451
Record Dates: First submitted 2017-11-10; First posted 2017-11-17 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Neoplasms; Radiotherapy Side Effect; Inflammation; Metabolism
Keywords: Head and neck cancer; Observational study; Three tertiary hospitals; Long-term follow-up; Survival; Immune response; Metabolomics
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries; Inflammation | interventions — Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample, tumor biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with head and neck cancer: All patients with newly diagnosed and untreated head and neck cancer. Exclusion criteria: previous treatment for malignant disorder except for skin cancer, severe alcohol abuse, psychiatric disorder, inability to understand Swedish
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — All patients will undergo radiotherapy or surgery, or combined modality treatment
  Other Names: Surgery

SUMMARY:
An estimated 1500 people in Sweden will annually be diagnosed with head and neck cancer (HNC). Five year survival is approximately 69%. Long-term sequelae are common and in particular nutritional problems and fatigue. Radiotherapy (RT) is the cornerstone of treatment, either as single modality treatment or combined modality treatment. RT can induce immune responses at the site of tumor. It has been demonstrated that RT can lead to a strong systemic immune response . We have previously shown that an increase of conventional measures of systemic immune response to RT varied significantly across individuals. We predict that local immune response plays a major role in the antitumor effect. We also predict that a strong systemic immune response contributes to malnutrition and influence on survival. And malnutrition may lead to a worse response to RT.

The overall aim of this multicenter observational longitudinal study is to prospectively identify immunological and metabolic variables that affect the outcome of HNC patients. We will systematically investigate the local and systemic immune response induced by RT as well as explore alterations in metabolite composition induced by disease and treatment through global metabolite profiling. A platform for studies on immuno-metabolic changes in HNC patients has been established in the Uppsala-Orebro and Northern regions. Approximately 370 patients per year are eligible. Findings in this study can have implications on the development of personalized therapy in patients with HNC. The long-term benefit of the study will be the identification of measures for improved patient surveillance in order to improve the general and nutritional outcomes.

DETAILED DESCRIPTION:
The incidence of head and neck cancer (HNC) has increased in Sweden during the last decades. Radiotherapy (RT) is a cornerstone of treatment either as single or combined modality treatment. There is emerging awareness that RT affects the immune system. For HNC patients treated with RT nutritional problems and fatigue are the most common long-term adverse effects. About 60% have advanced stage of disease at time of diagnosis. Recurrence as well as early death within two years is common.

Our hypothesis: there is a complex association between immune response, metabolic factors and survival.

The aim of this multicenter patient-centered observational longitudinal study is to prospectively identify immunological and nutritional/metabolic variables that affect the outcome of HNC patients. We will systematically investigate the local and systemic immune response induced by RT as well as explore alterations in metabolite composition induced by disease and treatment through global metabolite profiling (metabolomics). This highly biologically relevant data may be used to search for specific biomarkers of malnutrition, markers which would be of prognostic and/or diagnostic value. Moreover, analytically reliable data allows for a more comprehensive mechanistic understanding, as such, a particular focus lies in ensuring a high data quality. We have established a platform for a study on immuno-metabolic changes in HNC patients in the Uppsala-Orebro and Northern regions. Findings in this large-scale observational study can have implications on the development of personalized therapy in patients with HNC.

Survey of the field. There is restricted information on the importance of local and systemic immune response to RT in HNC patients. RT has systemic effects in addition to its local effects on tumors and surrounding tissue. Pro-inflammatory cytokines are activated by RT and have been associated with increased symptom burden in cancer treatment. Interleukin-6 (IL-6) is a potent inflammatory cytokine with diverse functions. In lung cancer mice xenograft studies irradiation has shown to induce an increase in IL-6 levels and migration of macrophages to the tumor tissue. An association between C-reactive protein (CRP) and IL-6 in plasma has been demonstrated in esophageal adenocarcinoma patients. Relapse-free patients are reported to have an increased proportion of Natural killer cells (NK-cells) in peripheral blood long-term after treatment. We have earlier followed a cohort of HNC patients during RT with repeated blood samples. high-sensitivity C-reactive protein (hCRP) increased during RT, and patients with the most pronounced weight loss had the greatest hCRP increase. Metabolic factors are reported to affect HNC patients in many ways. Severe malnutrition before treatment of HNC is reported to lead to increased mortality. In a secondary study in patients with oropharyngeal cancer (n = 357) we found that a high BMI gives significantly better 5-year survival than a low BMI. However, it is difficult to evaluate the results in the majority of nutritional studies in HNC patients because most prospective studies have included relatively few patients and many of the results obtained in retrospective studies have been conflicting. Patient's metabolic profile might work as a nutritional marker and be distinctly linked to nutritional status. The blood metabolome can be examined in detail in cancer patients to better identify different metabolic pathways. The nutritional status is strongly connected to the immune status. It is e.g. reported that L-arginine is crucial for the function of T-cell. As the immune system at the site of the tumor can inhibit cancer growth the local anti-tumorigenic immune status is important. Thus the nutritional status predicts the immune status and malnutrition is connected to a weaker immune response. It is unclear how the nutritional status is connected with the systemic immune status.

Research questions

1. The correlation between weight change and pro-inflammatory cytokines.
2. The correlation between weight change and immune response in tumour microenvironment.
3. Change of blood metabolome.
4. Change of Bioelectrical impedance analysis (BIA) measurements.
5. Change of fatty acid profile in blood.
6. Patient-reported outcome measure (PROM)
7. Patient-reported stress levels.
8. Return to work.
9. PROM and relation to treatment and overall survival.

Variables and measures All patients will be treated in accordance with local and national guidelines. Nutrient based local guidelines ensure that the patients receive nutritional support when needed. Baseline measurements will be taken before treatment starts, and follow-ups will take place at 4 and 7 weeks after start of treatment and at 3, 6, 12, and 24 months post treatment.

A Web-Based Patient Case Report Form (CRF) has been developed for a reliable, secure and easier data collection including the following variables:

Cancer-free survival, cancer-related death as well as death not related to cancer disease, interval between treatment and recurrence.

Explanatory variables:

1. Body Composition measured by BIA and validated against body composition measured by Dual-energy X-ray absorptiometry (DXA).
2. Characterization of immune profile in tumor tissue. Surgical biopsy of the tumor at the endoscopy for histopathological diagnosis and after RT when possible. Two methods will be applied to analyse the biopsies: 1) Multiplex tissue staining using the PerkinElmar Opal system which provides a quantitative and spatial composition of the immune cell infiltrates. 2) The RNA based Immunobiology Panel, which allows the measurement of the gene expression of hundreds of immune markers.
3. Immune profile in serum: analyzed with a multiplex assay using the Science for Life Laboratory (SciLife) platform.
4. Fatty acid profiling in serum with gas chromatography techniques.
5. Metabolomic parameters assessed with a multi-platform approach based on nuclear magnetic resonance (NMR) and high resolution mass spectrometry (HRMS) connected to the ultra-performance liquid chromatography (UPLC).
6. Body weight (kg) estimated 6 months before start of treatment, body weight registered at start of treatment and at all the follow-ups.

Questionnaires:

Nutritional follow-up with Patient Reported Outcome Measure Head and Neck Symptom Checklist (PROM - HNSC) (14). Quality of life (QoL) HNC specific questionnaire European Organization for Research and Treatment Quality of Life instrument (EORTC QLQ-H & N 35) (15). Hospital Anxiety and Depression Scale (HADS). Stress with questionnaire Perceived Stress Questionnaire (PSQ) (16).

Study design A prospective observational longitudinal study to elucidate all the research questions.

Estimated sample size About 1500 HNC patients are diagnosed annually in Sweden. The number of patients in this study before the exclusion criteria is approximately 370 patients/year.

Material: Patient selection - population, sample This multicenter study is a collaboration between the Uppsala-Orebro region and the Northern region. The patients are recruited at three university hospitals: Some of the patients are after treatment followed-up at their County Hospital. Inclusion criteria: curative treatment of patients with newly diagnosed HNC, and a World Health Organization (WHO) performance status of 0-2.

ELIGIBILITY:
Inclusion Criteria:

Patients with newly diagnosed head and neck cancer

Exclusion Criteria:

Previous treatment for malignant disease except for skin cancer, severe alcohol abuse, psychiatric disorder, inability to understand Swedish

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with head and neck cancer at the following three university hospitals:
  Uppsala University Hospital, Orebro University Hospital, Umea University Hospital
Sampling Method: Probability Sample
Enrollment: 522 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pro-inflammatory cytokines in serum | Change from baseline of pro-inflammatory cytokines in serum at 7 weeks
  IL-6
Pro-inflammatory cytokines in serum | Change from baseline of pro-inflammatory cytokines at 3 months
  IL-6
Pro-inflammatory cytokines in serum | Change from baseline of pro-inflammatory cytokines at 12 months
  IL-6

SECONDARY OUTCOMES:
Fatty acids in serum | Change from baseline of fatty acids at 7 weeks
  FA 14:0
Fatty acids in serum | Change from baseline of fatty acids at 3 months
  FA 14:0, FA 16:0, FA 18:0, FA 20:0
Fatty acids in serum | Change from baseline of fatty acids at 12 months
  FA 14:0
Weight | Change from baseline of weight to 7 weeks
  kilogram
Weight | Change from baseline of weight to 3 months
  kilogram
Weight | Change from baseline of weight at 12 months
  kilogram

CONTACTS AND LOCATIONS:
Overall Officials: Goran FE Laurell, Professor, Principal Investigator — Department of Otolaryngology, Head & Neck Surgery, Uppsala University Hospital
Locations (1):
- Department of Otolaryngology, Head & Neck Surgery, Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McBride WH, Chiang CS, Olson JL, Wang CC, Hong JH, Pajonk F, Dougherty GJ, Iwamoto KS, Pervan M, Liao YP. A sense of danger from radiation. Radiat Res. 2004 Jul;162(1):1-19. doi: 10.1667/rr3196. PMID 15222781
- [Background] Deorukhkar A, Krishnan S. Targeting inflammatory pathways for tumor radiosensitization. Biochem Pharmacol. 2010 Dec 15;80(12):1904-14. doi: 10.1016/j.bcp.2010.06.039. Epub 2010 Jun 30. PMID 20599771
- [Background] Wang C, Pu J, Yu H, Liu Y, Yan H, He Z, Feng X. A Dendritic Cell Vaccine Combined With Radiotherapy Activates the Specific Immune Response in Patients With Esophageal Cancer. J Immunother. 2017 Feb/Mar;40(2):71-76. doi: 10.1097/CJI.0000000000000155. PMID 28125513
- [Background] Hardikar S, Onstad L, Song X, Wilson AM, Montine TJ, Kratz M, Anderson GL, Blount PL, Reid BJ, White E, Vaughan TL. Inflammation and oxidative stress markers and esophageal adenocarcinoma incidence in a Barrett's esophagus cohort. Cancer Epidemiol Biomarkers Prev. 2014 Nov;23(11):2393-403. doi: 10.1158/1055-9965.EPI-14-0384. Epub 2014 Aug 8. PMID 25106775
- [Background] Bottcher A, Ostwald J, Guder E, Pau HW, Kramp B, Dommerich S. Distribution of circulating natural killer cells and T lymphocytes in head and neck squamous cell carcinoma. Auris Nasus Larynx. 2013 Apr;40(2):216-21. doi: 10.1016/j.anl.2012.07.004. Epub 2012 Jul 25. PMID 22835730
- [Background] Ehrsson YT, Hellstrom PM, Brismar K, Sharp L, Langius-Eklof A, Laurell G. Explorative study on the predictive value of systematic inflammatory and metabolic markers on weight loss in head and neck cancer patients undergoing radiotherapy. Support Care Cancer. 2010 Nov;18(11):1385-91. doi: 10.1007/s00520-009-0758-4. Epub 2009 Oct 15. PMID 19830461
- [Background] Datema FR, Ferrier MB, Baatenburg de Jong RJ. Impact of severe malnutrition on short-term mortality and overall survival in head and neck cancer. Oral Oncol. 2011 Sep;47(9):910-4. doi: 10.1016/j.oraloncology.2011.06.510. Epub 2011 Jul 28. PMID 21802345
- [Background] Capuano G, Grosso A, Gentile PC, Battista M, Bianciardi F, Di Palma A, Pavese I, Satta F, Tosti M, Palladino A, Coiro G, Di Palma M. Influence of weight loss on outcomes in patients with head and neck cancer undergoing concomitant chemoradiotherapy. Head Neck. 2008 Apr;30(4):503-8. doi: 10.1002/hed.20737. PMID 18098310
- [Background] Langius JA, Bakker S, Rietveld DH, Kruizenga HM, Langendijk JA, Weijs PJ, Leemans CR. Critical weight loss is a major prognostic indicator for disease-specific survival in patients with head and neck cancer receiving radiotherapy. Br J Cancer. 2013 Sep 3;109(5):1093-9. doi: 10.1038/bjc.2013.458. Epub 2013 Aug 8. PMID 23928661
- [Background] Huang S, Chong N, Lewis NE, Jia W, Xie G, Garmire LX. Novel personalized pathway-based metabolomics models reveal key metabolic pathways for breast cancer diagnosis. Genome Med. 2016 Mar 31;8(1):34. doi: 10.1186/s13073-016-0289-9. PMID 27036109
- [Background] Geiger R, Rieckmann JC, Wolf T, Basso C, Feng Y, Fuhrer T, Kogadeeva M, Picotti P, Meissner F, Mann M, Zamboni N, Sallusto F, Lanzavecchia A. L-Arginine Modulates T Cell Metabolism and Enhances Survival and Anti-tumor Activity. Cell. 2016 Oct 20;167(3):829-842.e13. doi: 10.1016/j.cell.2016.09.031. Epub 2016 Oct 13. PMID 27745970
- [Background] Schmidt KN, Olson K, Kubrak C, Parliament M, Ghosh S. Validation of the Head and Neck Patient Symptom Checklist as a nutrition impact symptom assessment tool for head and neck cancer patients. Support Care Cancer. 2013 Jan;21(1):27-34. doi: 10.1007/s00520-012-1483-y. Epub 2012 May 16. PMID 22588710
- [Background] Bjordal K, Hammerlid E, Ahlner-Elmqvist M, de Graeff A, Boysen M, Evensen JF, Biorklund A, de Leeuw JR, Fayers PM, Jannert M, Westin T, Kaasa S. Quality of life in head and neck cancer patients: validation of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-H&N35. J Clin Oncol. 1999 Mar;17(3):1008-19. doi: 10.1200/JCO.1999.17.3.1008. PMID 10071296
- [Derived] Tiblom Ehrsson Y, Einarsson S, Fransson P, Laurell G. Swedish Translation and Cultural Adaptation of the Head and Neck Patient Symptom Checklist: An Instrument to Screen for Nutrition Impact Symptoms in Clinical Practice and Research. West J Nurs Res. 2024 Oct;46(10):790-798. doi: 10.1177/01939459241274342. Epub 2024 Aug 24. PMID 39180372
- [Derived] Einarsson S, Bokstrom A, Laurell G, Tiblom Ehrsson Y. Mapping the impact of malnutrition as defined by the Global Leadership Initiative on Malnutrition and nutrition impact symptoms on the possibility of returning to work after treatment for head and neck cancer. Support Care Cancer. 2023 Dec 22;32(1):55. doi: 10.1007/s00520-023-08252-x. PMID 38133825
- [Derived] Granstrom B, Holmlund T, Laurell G, Fransson P, Tiblom Ehrsson Y. Addressing symptoms that affect patients' eating according to the Head and Neck Patient Symptom Checklist(c). Support Care Cancer. 2022 Jul;30(7):6163-6173. doi: 10.1007/s00520-022-07038-x. Epub 2022 Apr 15. PMID 35426524